CLINICAL TRIAL: NCT06831968
Title: Clinical Validation of a Predictive Test for Postpartum Depression
Acronym: PREVAIL
Status: Recruiting | Type: Observational
Sponsor: University of Virginia (Other)
Responsible Party: Principal Investigator, Jennifer L. Payne, Professor of Psychiatry and Neurobehavioral Sciences, University of Virginia
Other Study IDs: PR230933; HT94252410544 (Other Grant/Funding Number: Department of Defense)
Record Dates: First submitted 2025-01-17; First posted 2025-02-18 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-11

CONDITIONS: Postpartum Depression (PPD); Pregnancy
Keywords: Pregnancy; Postpartum Depression; Predictive Test; Blood Test; Third Trimester
MeSH Terms: conditions — Depression, Postpartum

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood and Saliva Samples
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | Unapproved Device: Yes

INTERVENTIONS:
Diagnostic Test: Enlighten — The primary analysis will examine the performance of the Enlighten Device by evaluating biomarker status results ("elevated risk" or "low risk") at the third trimester against depression symptoms outcome data collected by the 3 months postpartum time point.

SUMMARY:
The goal of this observational study is to develop a blood test that may be predictive of postpartum depression. This Blood test is investigational and not yet FDA approved. Participants will not receive the results of this blood test.

Up to 500 pregnant women will be recruited for the study from 2 sites. Participants must be age 18 or above with a singleton pregnancy and able to provide written consent in English.

The Objective of this Clinical Trial is to prospectively validate the Enlighten Device test by prospectively determining false/true positive and negative rates. Building off of this, an exploratory objective of this study is to examine clinical factors associated with false positive/negative rates.

This project will address the following Aim:

Aim 1: Prospective collection of true/false positive and negative PPD outcomes through 6 months postpartum.

Primary Hypothesis H1a: 80% or greater of pregnant women who develop PPD by 3 months after delivery will be determined to be Biomarker Positive by the Enlighten Device in T3.

Primary Hypothesis H1b: 10% or fewer of pregnant women who are determined to be Biomarker Negative by the Enlighten Device in T3 will develop PPD by 3 months after delivery.

Exploratory Aim 1: Investigation of clinical factors that may be associated with false positive and false negative rates, such as: medication use, stressful life events, and sociocultural context.

Participants will be screened during the second or third trimester and enrolled during the third trimester, before week 30 weeks of gestation. Participants may self- identify through study advertisements in participating clinics, social media outlets, and community outreach efforts. Enrolled participants will undergo blood collection during their 3rd trimester (~27-30 weeks, a standard pregnancy-related blood collection timepoint) for completion of the Enlighten Device test, the blood-based epigenetic biomarker test. Participants will then be interviewed at 2 weeks, 6 weeks, 3 months, and 6 months postpartum for the development of depression symptoms. They'll also complete a multitude of other outcome measures at each of these visits.

ELIGIBILITY:
Inclusion Criteria:

* subject must be pregnant (singleton pregnancy)
* <30 weeks' gestation, age 18 or above
* able to provide written consent in English

Exclusion Criteria:

* The study team and/or PI may exclude anyone deemed unsafe to participate in the protocol.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Up to 500 pregnant women, aged 18 years or above
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2025-03-20 (Actual); Primary Completion 2026-11-30 (Estimated); Study Completion 2028-07-31 (Estimated)

PRIMARY OUTCOMES:
Percentage of Participants with True/False Positive and Negative PPD Outcomes as Assessed by the Enlighten Device | 6 months postpartum
  PPD diagnosis will be confirmed by clinical evaluation using the Structured Clinical Interview for the DSM-5 Research Version (SCID-5-RV) and Edinburgh Postnatal Depression Scale (EPDS), at the time of enrollment and subsequent study visits. True positive/negative and false positive/negative classifications will be based on the Enlighten Device's biomarker threshold values in T3 (third trimester). Data will be aggregated as percentages and compared to clinical PPD diagnoses.
  Primary Hypothesis H1b: 10% or fewer of pregnant women who are determined to be Biomarker Negative by the Enlighten Device in T3 will develop PPD by 3 months after delivery.
  Exploratory Aim 1: Investigation of clinical factors that may be associated with false positive and false negative rates, such as: medication use, stressful life events, and sociocultural context.

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer L Payne, MD, Principal Investigator — University of Virginia; Andrea Cubitt, PhD, Principal Investigator — Dionysus Digital Health, Inc.
Locations (2):
- United States (2):
  - University of Virginia, Charlottesville, Virginia
  - Inova Health System, Falls Church, Virginia

IPD SHARING:
Plan to Share IPD: Yes
The investigators plan to share de-identified data with other researchers. Data shared will include demographic information, clinical data which will include SCID diagnosis, mental health surveys like EPDS, PASS, etc., sample analyses data.
Supporting Information: Study Protocol